CLINICAL TRIAL: NCT07251569
Title: The Effect of Mobile Application Deveoped for Postpartum Contraception Counseling on Contraception Method Choice and Use
Brief Title: The Effect of Mobile App Counseling on Postpartum Contraception Choices and Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burcu Dişli Oktar (Other)
Responsible Party: Sponsor-Investigator, Burcu Dişli Oktar, Research Assistant, PhD Student, RN, MSc, Istanbul University
Organization: Istanbul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023/76
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Contraception Use
Keywords: contraception; mobile application

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Other): Participants received no intervention and only received routine hospital postpartum care.
  Interventions: Other: Routine postpartum care
- Face-to-face counseling group (Active Comparator): Participants received contraception counseling and an educational booklet.
  Interventions: Behavioral: Face-to-face contraception counseling
- Mobile application counseling group (Experimental): Participants received contraceptive counseling through a mobile application developed as part of the study.
  Interventions: Behavioral: Contraceptive counseling via mobile application

INTERVENTIONS:
Other: Routine postpartum care — First Encounter: During the first five days postpartum, the postpartum woman was asked to complete the "Client Information Form" and "Contraceptive Information Form I." No intervention was performed. Postpartum women in this group received routine postpartum care offered to postpartum women in the hospital.
  First Follow-up: The client was called by phone at the sixth week postpartum. Breastfeeding status and whether she had initiated sexual intercourse were questioned. The "Contraceptive Information Form II" was completed by the researcher after being asked the client over the phone.
  Second Follow-up: The client was called again at the twelfth week postpartum. The "Follow-up Form" was completed by the researcher after being asked the client over the phone. At the end of the second follow-up, a general contraception counseling video was sent to the postpartum woman.
  Arms: Control Group
Behavioral: Face-to-face contraception counseling — First Encounter: During the first five days postpartum, the postpartum woman was asked to complete the "Client Information Form" and the "Contraceptive Information Form I." Sexuality during the postpartum period and the importance of contraception were then explained. Counseling on reproductive organ anatomy and general contraception was provided face-to-face, along with a booklet prepared as part of the research. At the end of the counseling, the booklet was given to the postpartum woman. She was told that she could review the booklet as often as she wished or needed.
  First Follow-Up: The client was contacted by phone at the sixth week postpartum. She was asked about her breastfeeding status and whether she had initiated sexual intercourse. The "Contraceptive Information Form II" was completed by the researcher over the phone.
  Second Follow-Up: The client was contacted again at the twelfth week postpartum. The "Follow-Up Form" was completed by the researcher over the phone.
  Arms: Face-to-face counseling group
Behavioral: Contraceptive counseling via mobile application — First Encounter: During the first five days postpartum, the postpartum woman was asked to complete the "Client Information Form" and "Contraceptive Information Form I." Information was provided about the importance of sexuality and contraception during the postpartum period. A postpartum contraception counseling mobile application was installed. The postpartum woman was asked to use the mobile application throughout the research period.
  First Follow-Up: The client was contacted by phone at the sixth week postpartum. She was asked about her mobile application use, breastfeeding status, and sexual intercourse status. The "Contraceptive Information Form II" was completed by phone. She was instructed to continue using the mobile application.
  Second Follow-Up: The client was contacted again at the twelfth week postpartum. She was asked about her mobile application use. The "Follow-Up Form" and "Mobile Application Evaluation Form" were completed by phone.
  Arms: Mobile application counseling group

SUMMARY:
The goal of this clinical trial is to determine the effect of a mobile application developed for postpartum contraception counseling on contraception method choice and use among postpartum women aged 18 and older. The main hypotheses it aims to answer are;

* H1: Among postpartum women, the use of highly effective contraceptive methods is higher in the group using a mobile application for contraception counseling compared to the group receiving face-to-face counseling.
* H2: Among postpartum women, the use of highly effective contraceptive methods is higher in the group using a mobile application for contraception counseling compared to the group receiving routine postpartum care.
* H3: Contraceptive method continuation and satisfaction are higher in the group using a mobile application for postpartum contraception counseling compared to the group receiving face-to-face counseling.
* H4: Contraceptive method continuation and satisfaction are higher in the group using a mobile application for postpartum contraception counseling compared to the group receiving routine postpartum care.

Researchers will compare three groups:

1. Group receiving contraception counseling via mobile app: Women in this group will have a postpartum contraception counseling mobile application installed on their phones and will use the application for 12 weeks.
2. Group receiving face-to-face contraception counseling: These women will receive face-to-face contraception counseling during the initial encounter, and an educational booklet will be provided at the end of the counseling session.
3. Control group: Women in this group will receive routine postpartum care. All groups will be followed up at three time points: the initial encounter, the first follow-up, and the second follow-up.

The initial encounter will be conducted face-to-face at the hospital within the first 5 days postpartum. The first follow-up will take place by phone at 6 weeks postpartum, and the second follow-up will be conducted by phone at 12 weeks postpartum.

DETAILED DESCRIPTION:
Reproductive and sexual health rights are part of fundamental individual rights. Every individual, regardless of gender, has the right to access quality reproductive health services and to decide freely whether or not to have children. Contraceptive counseling guides individuals to make their own informed decisions in line with these rights, without being directive. The postpartum period is a particularly suitable time to provide contraception counseling for planning future pregnancies. Furthermore, qualified counseling during this period helps prevent unintended pregnancies and contributes to the protection and improvement of maternal and child health. However, due to the short duration of hospital stays after childbirth, women may not feel ready to receive counseling during their stay. In addition, as mothers often prioritize the care of their newborns and older children, they may miss postpartum follow-up visits, resulting in contraception counseling not being delivered effectively.

International literature, including reports from the World Health Organization, has emphasized the inadequate provision of contraception counseling during the postpartum period and highlighted the development of mobile applications to address this issue. These applications assist individuals in choosing safe, effective, and appropriate contraceptive methods, enabling them to easily manage and monitor their reproductive health. Moreover, mobile applications contribute to national health systems by reducing costs and improving access to contraception counseling services for individuals living in rural or underserved areas, allowing access anytime and anywhere.

This study aims to develop a mobile application specifically designed for postpartum contraception counseling and to determine its effect on postpartum women's contraceptive method choice and continued use.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Being within the first 5 days postpartum
* Having a healthy newborn
* Not having received fertility treatment for the last pregnancy
* Not having undergone tubal ligation during delivery
* Owning a smartphone
* Being able to use a mobile application
* Having internet access
* Being able to speak, read, and write in Turkish

Exclusion Criteria:

* Having previously received contraceptive counseling
* Discontinuing the use of the mobile application
* Not participating in follow-up visits
* Not volunteering to participate in the study
* Having a diagnosed psychiatric disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Choice of contraceptive method and its effectiveness level | First Encounter (in the first 5 days postpartum) First Follow-Up (in the 6th week postpartum) Second Follow-Up (in the 12th week postpartum)
  The chosen contraceptive method and its effectiveness were categorically assessed using a "Client Information Form" at the first visit, a "Contraceptive Information Form II" at the first follow-up, and a "Follow-up Form" at the second follow-up. All three forms were developed by the researchers based on the relevant literature. The effectiveness of the contraceptive methods was determined according to the World Health Organization's estimates of unintended pregnancy rates during the first year of typical use. Methods with unintended pregnancy rates of less than 10% in the first year of typical use were classified as highly effective, whereas methods with rates of 10% or higher were classified as less effective.
Level of satisfaction with the chosen contraceptive method | Second Follow-Up (at the 12th postpartum week)
  Satisfaction with the chosen contraceptive method was measured numerically at the second follow-up using a question on the "Follow-up Form," scored from 1 to 10. A score of 1 means "I am not satisfied at all," and a score of 10 means "I am very satisfied." A higher score indicates higher satisfaction.
Status of continuing the chosen contraceptive method | Second Follow-Up (at the 12th postpartum week)
  Continuity with the chosen contraceptive method was measured categorically at the second follow-up using the "Follow-up Form" developed by the researchers based on literature.

SECONDARY OUTCOMES:
Knowledge status regarding contraceptive methods | First Encounter (in the first 5 days postpartum) First Follow-Up (in the 6th week postpartum) Second Follow-Up (in the 12th week postpartum)
  The knowledge status regarding contraceptive methods was categorically assessed using the "Contraceptive Information Form I" at the first visit, the "Contraceptive Information Form II" at the first follow-up, and the "Follow-up Form" at the second follow-up. These forms were developed by the researchers based on the relevant literature. The forms include questions about which contraceptive methods the participants had previously heard of, which methods they had knowledge about, and their understanding of the characteristics of contraceptive methods.
Mobile Application Evaluation Form Results | Second Follow-Up (in the 12th week postpartum)
  The Mobile Application Evaluation Form was developed by researchers based on literature. The forms evaluate the content, visual appearance, usability, and features of the mobile application developed for the research, using 12 items. The first 11 items are evaluated with "Yes" or "No" responses, while the 12th item is open-ended.

OTHER OUTCOMES:
Assessment of Sociodemographic, Obstetric, and Gynecological Characteristics | First Encounter (in the first 5 days postpartum)
  Sociodemographic, obstetric, and gynecological characteristics were assessed numerically and categorically at the first encounter using a "Client Information Form" developed by the researchers based on literature. Data included in this form include age, age at first menstruation, menstrual duration, frequency, number of pregnancies, number of vaginal births, number of cesarean sections, etc., which are assessed numerically; and marital status, education level, income status, social security status, smoking status, menstrual cycle patterns, etc., which are assessed categorically.

CONTACTS AND LOCATIONS:
Locations (1):
- Esenler Maternity and Child Diseases Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the absence of participant consent for external data sharing and institutional policies that restrict the release of raw data.

REFERENCES:
- [Background] Berrami H, Serhier Z, Jallal M, Bennani Othmani M. Mobile Applications for Family Planning. Stud Health Technol Inform. 2023 Oct 20;309:300-301. doi: 10.3233/SHTI230803. PMID 37869864
- [Result] Sze YY, Berendes S, Russel S, Bellam L, Smith C, Cameron S, Free CJ. A systematic review of randomised controlled trials of the effects of digital health interventions on postpartum contraception use. BMJ Sex Reprod Health. 2023 Jan;49(1):50-59. doi: 10.1136/bmjsrh-2022-201468. Epub 2022 Oct 28. PMID 36307185
- [Result] Cherie N, Wordofa MA, Debelew GT. Effectiveness of an Interactive Mobile Health Intervention (IMHI) to enhance the adoption of modern contraceptive methods during the early postpartum period among women in Northeast Ethiopia: A cluster Randomized Controlled Trial (RCT). PLoS One. 2024 Nov 14;19(11):e0310124. doi: 10.1371/journal.pone.0310124. eCollection 2024. PMID 39541340
- [Result] Dev R, Woods NF, Unger JA, Kinuthia J, Matemo D, Farid S, Begnel ER, Kohler P, Drake AL. Acceptability, feasibility and utility of a Mobile health family planning decision aid for postpartum women in Kenya. Reprod Health. 2019 Jul 8;16(1):97. doi: 10.1186/s12978-019-0767-9. PMID 31286989
- [Result] Sonalkar S, Maya E, Adanu R, Samba A, Mumuni K, McAllister A, Fishman J, Schurr D, Schreiber CA, Kolev S, Doe R, Eluned Gaffield M. Pilot monitoring and evaluation of the WHO postpartum family planning compendium mobile application: An in-depth, qualitative study. Int J Gynaecol Obstet. 2021 Jun;153(3):508-513. doi: 10.1002/ijgo.13631. Epub 2021 Mar 2. PMID 33513267